CLINICAL TRIAL: NCT03054181
Title: Facilitated Immunoglobulin Administration Registry and Outcomes Study
Brief Title: Facilitated Immunoglobulin Administration Registry and Outcomes Study (FIGARO)
Acronym: FIGARO
Status: Completed | Type: Observational
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: FIGARO
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2022-03

CONDITIONS: Primary Immunodeficiency; Secondary Immune Deficiency
Keywords: Observational; Infection; Utilisation; Safety; Tolerability; Infusion; chronic
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Infections; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HyQvia: Recombinant human hyaluronidase and normal immunoglobulin 10%
  Interventions: Biological: HyQvia

INTERVENTIONS:
Biological: HyQvia
  Other Names: Recombinant human hyaluronidase and normal immunoglobulin 10%

SUMMARY:
Long-term observational study on the utilisation and outcomes of HyQvia (a product consisting of recombinant human hyaluronidase and a human normal immunoglobulin 10% solution) under everyday clinical practice conditions.

DETAILED DESCRIPTION:
Recombinant hyaluronidase is an established therapeutic principle to facilitate the infusion of large volumes of fluids subcutaneously (e.g. Ringer solution and antibodies such as IG, rituximab, trastuzumab).

HyQvia is a product consisting of recombinant human hyaluronidase (rHuPH20, Hylenex®), and a human normal immunoglobulin (IG). The subcutaneous (SC) IG is a 10% solution prepared from human plasma consisting of at least 98% immunoglobulin G, which contains a broad spectrum of antibodies.

The two components are packaged together as a dual vial unit: IG provides the therapeutic effect and the recombinant human hyaluronidase facilitates the dispersion, which alters the kinetics of absorption and increases the bioavailability of the IG.

HyQvia is marketed in the European Union (EU) since July 2013 and in the USA since September 2014. In the EU, HyQvia is indicated as replacement therapy in patients of all age groups in primary immunodeficiency syndromes (PID), and in myeloma or chronic lymphocytic leukaemia with severe secondary hypogammaglobulinaemia and recurrent infections (secondary immunodeficiency syndromes, SID), as well as hypogammaglobulinaemia and pre- and post-allogeneic hematopoietic stem cell transplantation.

HyQvia was investigated in one pivotal study lasting over a year, involving 89 patients with PID who had already had treatment with human normal IG for at least three months. The number of acute serious bacterial infections (SBI) as main efficacy outcomes was 0.025 per year. This was below the FDA predefined number needed to show efficacy (SBI rate <1.0 per subject per year at the 0.01 level of significance), and was similar to that seen with other licensed human normal IG products. In the pivotal study and its extension, 188 patient years under HyQvia treatment have been documented. HyQvia was efficacious, safe, and bioequivalent to intravenous IG at the same administration intervals, but it caused fewer systemic reactions. Tolerability was good despite high infusion volumes and rates. There are no preclinical data that suggest an increased risk of mutagenicity, teratogenicity, fertility or neuronal development.

The most current and comprehensive data on real-life utilisation and outcomes of various IgG preparations is available from the German SIGNS registry. This registry confirmed the effectiveness of IgG substitution or treatment in terms of reduction of infections (PID and SID), as well as stabilization or improvement of the clinical condition in neurological and autoimmune diseases. In a cohort of 24 PID and SID patients on HyQvia in the German SIGNS study, the preparation was well tolerated and treatment satisfaction was high. In other countries, data on the utilisation and outcomes of HyQvia under clinical practice conditions are sparse or completely missing.

The present study aims to fill these gaps and to provide a detailed and complete description of the utilisation of under everyday clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient has received/will receive at least 1 HyQvia infusion for PID or SID
* Patient has an indication for chronic immunoglobulin treatment
* Patient is likely available for long-term documentation
* Patient provides informed consent for documentation

Exclusion Criteria:

* No explicit exclusion criteria apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary (PID) or secondary immunodeficiencies (SID)
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Utilisation in terms of dose and dosing interval | up to 3 years
  mean monthly dose

SECONDARY OUTCOMES:
Adverse events | up to 3 years
  Incidence and type
Concomitant diseases | up to 3 years
mean immunoglobulin trough level | up to 3 years
  after HyQvia infusion
Number of participants with treatment-related adverse events | up to 3 years
  Acute bacterial infections; overall infections
Number of training session | up to 3 years
  about appropriate self-infusion
Number of days in hospital | up to 3 years
Number of days in rehabilitation clinic | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Borte, MD, PhD, Principal Investigator — Fachbereich Pädiatrische Rheumatologie, Immunologie und Infektiologie am Klinikum St. Georg Leipzig; David Pittrow, MD, Study Director — GWT-TUD GmbH, Dresden, Germany; Isabelle Quinti, MD, Study Chair — Sapienza University Rome, Italy; Leif Hanitsch, MD, Study Chair — Charité Berlin, Germany; Nizar Mahlaoui, MD, Study Chair — University Hospital, Paris, France
Locations (4):
- University Hospital, Paris, France
- Germany (2):
  - Charité, Berlin
  - Hospital for Children and Adolescents, St. Georg Hospital, Academic Teaching Hospital, Leipzig
- La Sapienza University, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Borte M, Hanitsch LG, Mahlaoui N, Fasshauer M, Huscher D, Speletas M, Dimou M, Kamieniak M, Hermann C, Pittrow D, Milito C. Facilitated Subcutaneous Immunoglobulin Treatment in Patients with Immunodeficiencies: the FIGARO Study. J Clin Immunol. 2023 Aug;43(6):1259-1271. doi: 10.1007/s10875-023-01470-2. Epub 2023 Apr 10. PMID 37036560